CLINICAL TRIAL: NCT06457568
Title: Validation of the CONTEC08C Oscillometric Blood Pressure Monitor in General Population According to the AAMI/ESH/ISO Universal Standard (ISO 81060-2:2018)
Brief Title: Validation Study of CONTEC08C Electronic Sphygmomanometer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Lou ying, MD, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-ZX082
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONTEC08C and mercury sphygmomanometer (Experimental): Blood Pressure Measurement with the CONTEC08C Oscillometric Sphygmomanometer (CONTEC08C) and with Mercury Sphygmomanometer
  Interventions: Diagnostic Test: Blood pressure measurement

INTERVENTIONS:
Diagnostic Test: Blood pressure measurement — The blood pressure measurement was taken simultaneously by two observers using mercury sphygmomanometer and by a supervisor using the tested device, CONTEC08C.

SUMMARY:
The purpose of this study is to assess the accuracy of the CONTEC08C automated oscillometric upper-arm sphygmomanometer in the general population for clinical use according to the Association for the Advancement of Medical Instrumentation/European Society of Hypertension /International Organization for Standardization (AAMI/ESH/ISO) Universal Standard (ISO 81060-2:2018).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 12 to 79 years
* Subjects voluntarily participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

* Subjects with cardiac arrhythmias;
* Pregnancy;
* Poor quality Korotkoff sounds;
* Subject with an arm injury incompatible with the use of a cuff-based sphygmomanometer;
* Other conditions that the investigator considers ineligible for clinical trial.

Ages: 12 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-25 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure measurement data | 30mintues
  Systolic Blood Pressure and Diastolic Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lou, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Sciences，Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No